CLINICAL TRIAL: NCT05630300
Title: Assessing the Feasibility and Usability of Implementing Professional Use and Self-administered COVID-19 Antigen RDTs in Uganda
Brief Title: Feasibility and Usability of COVID-19 Antigen RDTs in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RES-00378
Record Dates: First submitted 2022-11-21; First posted 2022-11-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facility-based Ag-RDT COVID-19 testing - reactive (Experimental): Out-patient department patients who utilized a COVID-19 Ag-RDT professional-use test in an OPD clinical setting with reactive test result
  Interventions: Diagnostic Test: PMC Sure Status COVID-19 Antigen Test
- Facility-based Ag-RDT COVID-19 testing - non-reactive (Experimental): Out-patient department patients who utilized a COVID-19 Ag-RDT professional-use test in an OPD clinical setting with non-reactive test result
  Interventions: Diagnostic Test: PMC Sure Status COVID-19 Antigen Test
- COVID-19 Ag-RDT self-testing - agree to self-test (Experimental): Participants who receive and take a COVID-19 Ag-RDT self-test (female sex workers, Boda boda drivers, household contacts)
  Interventions: Diagnostic Test: Acon Flowflex COVID-19 Antigen Home Test
- COVID-19 Ag-RDT self-testing - refuse to self-test (No Intervention): Participants who receive but refuse to take a COVID-19 Ag-RDT self-test (female sex workers, Boda boda drivers, household contacts)

INTERVENTIONS:
Diagnostic Test: PMC Sure Status COVID-19 Antigen Test — COVID-19 professional use kit in out-patient departments
  Arms: Facility-based Ag-RDT COVID-19 testing - non-reactive; Facility-based Ag-RDT COVID-19 testing - reactive
Diagnostic Test: Acon Flowflex COVID-19 Antigen Home Test — COVID-19 self-test kits
  Arms: COVID-19 Ag-RDT self-testing - agree to self-test

SUMMARY:
This study will assess the feasibility and usability of COVID-19 professional and self-administered Antigen-Rapid Diagnostic Tests (Ag-RDTs) through health facility outpatient services and community settings in Kampala and Luwero districts in Uganda.

There are two components to this study:

1. Facility-based COVID-19 Ag-RDT professional use testing which will include people seeking care at outpatient departments and household contacts of index participants diagnosed at outpatient departments in four health facilities in Kampala and Luwero districts.
2. Community-based COVID-19 Ag-RDT self-testing which will include at-risk populations such as female sex workers (FSW) and Boda boda drivers (motorcyclists) at points of mass throughfare in Kampala and Luwero districts.

Key outcomes target the implementation's success, demand, and usability of professional and self-administered Ag-RDTs.

DETAILED DESCRIPTION:
This study seeks to understand the feasibility and usability of COVID-19 Ag-RDT self-tests among Boda boda drivers and FSWs in community-based settings in two districts of Uganda. Ag-RDT COVID-19 professional use tests will also be assessed, among patients soliciting OPD services in health facilities, to support public-sector screening when qRT-PCR testing services are limited or unavailable. Feasibility for the purposes of this intervention refers to core factors affecting implementation success (i.e., barriers, facilitators, user preferences, and acceptability of Ag-RDT use and implementation) and demand (the measure of actual use of professional and self-administered Ag-RDTs in the population). Usability is defined as the extent to which FSWs, Boda boda drivers, and OPD patients, and household contacts of OPD patients self-report their comfort with performing critical self-testing procedures (sample collection, sample processing, and results interpretation) autonomously.

Primary Research Objective

• To assess the feasibility of using professional and self-administered COVID-19 Ag-RDTs in facility OPD and community settings in Uganda.

Secondary Research Objective • Determine usability of Ag-RDT COVID-19 self-tests among FSWs, Boda boda drivers, OPD patients, and household contacts of OPD patients.

Primary outcomes: Feasibility of professional and self-administered COVID-19 Ag-RDT use.

* Implementation success. Number of people who report COVID 19 self-testing and professional COVID 19 testing acceptable and preferred.
* Demand. Proportion of COVID-19 OPD cases identified via professional use testing who accept to take self-testing kits for their contacts.
* Demand. Proportion of FSWs, Boda boda drivers, and household contacts who use Ag-RDT COVID-19 self-tests and report their findings.

Secondary outcomes: Usability of Ag-RDT self-administered tests.

• Usability. Proportion of assisted self-testers compared to unassisted self-testers who self-report that they feel comfortable using the test and return the results, stratified by population group (OPD patients, household contacts of OPD patients, FSWs, and Boda boda drivers).

ELIGIBILITY:
OPD patients (index cases) for professional use testing

Inclusion Criteria:

* 18 years of age or older or below 18 years and meets the qualification of an emancipated minor (heads a family, takes care of his/herself, pregnant/has children, cohabiting or married).
* Exhibits signs and symptoms of a COVID-19 infection.
* Positive screening result for COVID-19 infection using -Ag-RDT self-test or Ag-RDT professional-use test.
* Willing and able to provide informed consent to participate and comply with study requirements.

Exclusion Criteria:

* Any study site employees who are involved in the protocol or may have access to study-related data.
* Treating clinician deems inappropriate to enroll.
* Those who do not have a telephone contact to report results and be interviewed on phone.

Household contacts of OPD patients for self-testing

Inclusion Criteria:

* 18 years of age or older or below 18 years and meets the qualification of an emancipated minor (heads a family, takes care of his/herself, pregnant/has children, cohabiting or married).
* Exposure to COVID-19 (i.e., being within 6ft/1 meter of the index case for more than 15 minutes or physical contact with the index case within the 2 days before symptom onset of the confirmed COVID-19 case (index case).
* Willing and able to provide informed consent.

Exclusion Criteria

* Contraindication to nasal swab.
* Had a nasopharyngeal swab in the last 8 hours.
* Any study site employees who are involved in the protocol or may have access to study-related data.
* Already enrolled in this study.

Community-based self-testing participants (FSWs and Boda boda drivers)

Inclusion criteria:

* 18 years of age or older or below 18 years and meets the qualification of an emancipated minor (heads a family, takes care of his/herself, pregnant/has children, cohabiting or married).
* Must identify as a FSW or Boda boda driver.
* Ability to provide informed consent.
* Must be a resident or working in Kampala or Luwero districts.

Exclusion Criteria:

* Unwilling or unable to provide informed consent.
* Not a part of the population group outlined above.
* Has no cell phone to convey results and for interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Implementation success | 6 months
  Proportion of focus group discussion responses on the barriers, facilitators, user preferences, and acceptability to offering COVID-19 Ag-RDT professional and self-administered kits in health facilities and community settings through thematic analysis.
Demand - OPD | 6 months
  Proportion of COVID-19 OPD cases identified via professional use testing who accept self-testing kits for their contacts.
Demand - Community | 6 months
  Proportion of FSWs, Boda boda drivers, and household contacts who use Ag-RDT COVID-19 self-tests and report their results.

SECONDARY OUTCOMES:
Usability | 6 months
  Proportion of assisted self-testers compared to unassisted self-testers who self-report their comfort with correctly using the test and return the results, stratified by population group (OPD patients, household contacts of OPD patients, FSWs, and Boda boda drivers).

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Green, Principal Investigator — PATH
Locations (4):
- Uganda (4):
  - Kisenyi Health Center IV, Kampala, Central Region
  - Kiswa Health Center III, Kampala, Central Region
  - Katikamu Health Center III, Luwero, Central Region
  - Luwero Hospital, Luwero, Central Region

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share any individual participant data, as study data will be aggregated into the study database for analysis and further dissemination of results.